CLINICAL TRIAL: NCT04642573
Title: The Metabolic Characteristics in Sublobar Areas of Pharmacoresistant Epilepsy Based on FDG-PET Study
Brief Title: The Metabolic Characteristics in Sublobar Areas of PRE Based on FDG-PET Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-743
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Interictal FDG-PET Hypometabolism Patterns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non interventional — non interventional

SUMMARY:
Epilepsy is a chronic brain disease that is caused by various factors and characterized by recurrent, episodic and temporary central nervous system dysfunction. In the past few decades, despite the continuous development of antiepileptic drugs, there are still 20%-30% patients with epilepsy progressing to pharmacoresistant epilepsy (PRE), which leads to a significant increase in the morbidity and mortality of epilepsy. For those fraction of PRE, surgical treatment may be the only possible way to cure epilepsy. Accurate presurgical evaluation play an important role in making surgery decision and defining surgical extent and achieve better surgical outcome. Imaging, especially interictal fluorine-18-fluorodeoxyglucose-positron emission tomography (FDG-PET) is widely used in preoperative evaluation, which is of great significance in the detection of epileptogenic foci. Previous studies on FDG-PET have found that FDG-PET has a wide range of hypometabolism inpatients of PRE varying from different epileptic origins. Therefore, exploring the characteristics of glucose metabolism originating in different brain areas of resistant epilepsy can help to better interpret the results of FDG-PET and guide the preoperative localization of such patiens and better understand the potential mechanism of seizure propagation in PRE.

ELIGIBILITY:
Inclusion Criteria: (a) Pharmacoresistant Epilepsy may be defined by International League Against Epilepsy (ILAE）as failure of adequate trials of two tolerated and appropriately chosen and used AED schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom (judged by two epileptologists); (b) conventional MRI negative or nonspecific abnormalities; and (c) detailed information of long-term video-EEG, FDG-PET, high resolution MRI (HR-MRI) and neuropsychological assessment were acquired, (d) focal epilepsy defined by combining clinical, electrophysical and neuroimaging.

Exclusion Criteria: (a) generalized or multifocal epilepsy or the patient's electroclinical features were inconsistent with pharmacoresistant epilepsy; (b) idiopathic focal epilepsy; and (c) unsatisfactory imaging quality.

-

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We prospectively recruited 100 consecutive patients with pharmacoresistant epilepsy at our epilepsy center since Nov 2020. All the patients should have agreed to sign an informed consent.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
hypometabolic patterns for each patient group comparing with control group | 1-3months
  Due to the different epileptogenic zones in each group, the hypometabolic patterns should be different

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided